CLINICAL TRIAL: NCT02744235
Title: Sensitivity and Specificity of Mainstream Sleep Tracking Devices Compared to Polysomnography
Brief Title: Mainstream Sleep Tracking Devices vs Polysomnography
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to move forward due to funding
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-00071
Record Dates: First submitted 2016-04-13; First posted 2016-04-20 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Severe Sleep Apnea; Severe Insomnia; Epileptiform Activity
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients undergoing Polysomnography (Other)
  Interventions: Device: Polysomnography Data; Device: Jawbone UP®; Device: Fitbit Charge ®

INTERVENTIONS:
Device: Polysomnography Data
Device: Jawbone UP®
Device: Fitbit Charge ®

SUMMARY:
The purpose of this study is to compare two popular portable sleep monitoring devices-the Fitbit Charge®, Jawbone UP®, and SleepTime smartphone app-to the "gold standard" Polysomnography (PSG). Parameters that will be analyzed include sleep onset latency, sleep efficiency, and sleep staging. Specifically, this study will investigate the validity of the Jawbone UP®, Fitbit Charge®, and SleepTime app in detecting sleep and wakefulness in comparison to conventional Polysomnography (PSG).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Polysomnography

Exclusion Criteria:

* severe sleep apnea
* severe insomnia with less than two hours of sleep per night
* epileptiform activity
* electrical status epilepticus of sleep

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Time it takes subject to fall asleep | Up to 3 Months
Number of Minutes of Sleep | Up to 3 Months
Number of Arousals | Up to 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Alcibiades Rodriguez, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States